CLINICAL TRIAL: NCT02678247
Title: Functional Performance Evaluation of the Northwestern University Flexible Sub-Ischial Vacuum (NU-FlexSIV) Socket for Persons With Transfemoral Amputation
Brief Title: Functional Performance Evaluation of NU-FlexSIV Socket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Jesse Brown VA Medical Center (U.S. Federal Agency); Scheck and Siress (Industry)
Responsible Party: Principal Investigator, Stefania Fatone, PhD, BPO(Hons), Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-15-1-0708
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Amputation; Artificial Limbs
Keywords: prosthesis; prosthetic socket; transfemoral amputation; socket comfort; gait biomechanics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NU-FlexSIV Socket (Active Comparator): The Northwestern University Flexible Sub-Ischial Vacuum Socket is a novel socket design for transfemoral amputees.
  Interventions: Device: Northwestern University Flexible Sub-Ischial Vacuum Socket; Device: Ischial Containment Socket
- IC Socket (Active Comparator): The Ischial Containment Socket is the standard of care socket design for transfemoral amputees.
  Interventions: Device: Northwestern University Flexible Sub-Ischial Vacuum Socket; Device: Ischial Containment Socket

INTERVENTIONS:
Device: Northwestern University Flexible Sub-Ischial Vacuum Socket — NU-FlexSIV sockets have lower proximal trim lines, do not impinge on the pelvis, are highly flexible so as to allow better comfort during sitting and when muscles move within the socket during activity, and are held securely to the residual limb by suction from a vacuum pump and from compression exerted by the deliberately undersized liner and socket.
  Other Names: NU-FlexSIV Socket
Device: Ischial Containment Socket — Ischial Containment (IC) sockets are more rigid and have a narrower medio-lateral dimension than anterior-posterior dimension. The socket encapsulates the ischium, ischial ramus and greater trochanter, limiting hip range of motion and comfort.
  Other Names: IC Socket

SUMMARY:
The overall objective of this study is to provide a more comfortable and functional prosthetic socket for persons with transfemoral amputation that will ultimately improve their quality of life.

DETAILED DESCRIPTION:
The proposed clinical trial will be an assessor-blinded prospective randomized cross-over trial wherein participants with unilateral transfemoral amputation will be randomized to using one of two socket conditions (i.e., sub-ischial or ischial containment) before crossing over to the other socket condition. Random allocation (computer-generated) utilizing blocks of random size will be used to assign the initial treatment condition. The trial will be balanced such that all subjects will receive all treatments (i.e., both socket conditions) and that all subjects will participate for the same number of periods (i.e., two). While a washout period is not strictly necessary, it is effectively included as subjects will need to transition back to their usual, pre-study socket/prosthesis while the second test socket is fabricated.

Allocation of intervention will be concealed from the investigators until after a subject is enrolled. The starting socket design will be enclosed in sequentially numbered, opaque, sealed envelopes. Envelopes will be opened sequentially and only after the participant's name and other details are written on the appropriate envelope.

Blinding of prosthetic interventions is challenging given that they are devices that must be custom-fabricated and donned each day by the subject. Hence, for this study only the assessor will be blinded. The blinded assessor will be responsible for administration of the clinical performance and patient-reported measures as well as processing of motion analysis data.

ELIGIBILITY:
Inclusion Criteria:

* unilateral transfemoral amputation
* have used a prosthesis for two or more years
* have a residual limb that is stable in volume and free from wounds
* be physically fit enough to participate in the performance tests (Medicare Functional Classification Level K3 or K4)
* have no previous experience of the sub-ischial socket
* able to complete all visits for the duration of the protocol

Exclusion Criteria:

* have a residual limb femur of less than 5-inches
* co-morbidities that affect function, including neurologic abnormalities (e.g. neuropathic pain that would interfere with the study)
* do not speak and read English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fatone, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Jesse Brown VA Medical Center Motion Analysis Research Laboratory, Chicago, Illinois
  - Northwestern University Prosthetics-Orthotics Center, Chicago, Illinois
  - Scheck and Siress Prosthetics Orthotics, Oakbrook Terrace, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Upon request, the PI will share de-identified data and outcomes. If the requests are excessive, data will be made available via a link on the Northwestern University Prosthetics-Orthotics Center (NUPOC) website.
Time Frame: Once results are published.
Access Criteria: Upon request, the PI will share de-identified data and outcomes. If the requests are excessive, data will be made available via a link on the Northwestern University Prosthetics-Orthotics Center (NUPOC) website.
URL: https://www.nupoc.northwestern.edu/research/projects/lowerlimb/FunctionalPerfEvalNUFlexSIV.html

REFERENCES:
- [Derived] Fatone S, Stine R, Caldwell R, Angelico J, Gard SA, Oros M, Major MJ. Comparison of Ischial Containment and Subischial Sockets Effect on Gait Biomechanics in People With Transfemoral Amputation: A Randomized Crossover Trial. Arch Phys Med Rehabil. 2022 Aug;103(8):1515-1523. doi: 10.1016/j.apmr.2022.02.013. Epub 2022 Mar 13. PMID 35296398
- [Derived] Fatone S, Caldwell R, Angelico J, Stine R, Kim KY, Gard S, Oros M. Comparison of Ischial Containment and Subischial Sockets on Comfort, Function, Quality of Life, and Satisfaction With Device in Persons With Unilateral Transfemoral Amputation: A Randomized Crossover Trial. Arch Phys Med Rehabil. 2021 Nov;102(11):2063-2073.e2. doi: 10.1016/j.apmr.2021.05.016. Epub 2021 Jun 29. PMID 34214499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 2016 and May 2019. Subjects were recruited and sockets fit and fabricated at local prosthetic clinical care facilities. Data were collected in an academic research lab.
Pre-assignment Details: 30 subjects were randomized.
Groups:
- Ischial Containment Socket Then NU-FlexSIV Socket: Participants first received the Ischial Containment Socket which they wore for 7 weeks, then they received the NU-FlexSIV Socket which they wore for 7 weeks.
- NU-FlexSIV Socket Then Ischial Containment Socket: Participants first received the NU-FlexSIV Socket which they wore for 7 weeks, then they received the Ischial Containment Socket which they wore for 7 weeks.
Period: First Intervention (7 Weeks)
Arm/Group | Ischial Containment Socket Then NU-FlexSIV Socket | NU-FlexSIV Socket Then Ischial Containment Socket
Started | 15 | 15
Completed | 13 | 11
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 1 | 0
Period: Second Intervention (7 Weeks)
Arm/Group | Ischial Containment Socket Then NU-FlexSIV Socket | NU-FlexSIV Socket Then Ischial Containment Socket
Started | 14 (One subject crossed over despite not completing all data collection time points for the preceding socket.) | 11
Completed | 10 | 9
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ischial Containment Socket Then NU-FlexSIV Socket: Participants wore the Ischial Containment Socket for 7 weeks then wore the NU-FlexSIV Socket for 7 weeks.
- NU-FlexSIV Socket Then Ischial Containment Socket: Participants wore the NU-FlexSIV Socket for 7 weeks then wore the Ischial Containment Socket for 7 weeks.
- Total: Total of all reporting groups
Arm/Group | Ischial Containment Socket Then NU-FlexSIV Socket | NU-FlexSIV Socket Then Ischial Containment Socket | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data missing for subjects who withdrew before first data collection session.
  years
    number analyzed (Participants) | 14 | 11 | 25
    (all) | 50.6 (13.7) | 39.9 (11.6) | 45.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 14 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Time Since Amputation [Mean (Standard Deviation); unit: years] — Population: Data missing for subjects who withdrew before first data collection session.
  years
    number analyzed (Participants) | 14 | 11 | 25
    (all) | 27.6 (17.1) | 17.6 (12.7) | 23.2 (15.8)
Cause of Amputation [Count of Participants; unit: Participants]
  Trauma | 9 | 6 | 15
  Cancer | 4 | 3 | 7
  Vascular | 1 | 1 | 2
  Infection | 0 | 1 | 1
  Unknown | 1 | 4 | 5
K-Level Classification [Count of Participants; unit: Participants] — Rating system used by Medicare to indicate a person's rehabilitation potential. Rating from 0 to 4 indicates a person's potential to use a prosthetic device. K0: no ability/potential. K1: household ambulator. K2: limited community ambulator. K3: community ambulator. K4: exceeds basic ambulation skills.
  Participants
    K3 | 4 | 3 | 7
    K4 | 11 | 12 | 23
Amputee Mobility Predictor with Prosthesis [Mean (Standard Deviation); unit: score: 0-47] — A 21-item performance-based measure of ambulatory potential with a lower limb prosthesis. Scored from 0 to 47, with higher scores indicating better ambulatory ability with prosthesis. Population: Data missing for subjects who withdrew before first data collection session.
  score: 0-47
    number analyzed (Participants) | 14 | 11 | 25
    (all) | 43.2 (1.8) | 42.1 (3.2) | 42.7 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Socket Comfort Score (SCS) Between IC Socket and NU-FlexSIV Sockets at 7 Weeks.
Description: Socket comfort was assessed after each socket was worn for 7 weeks. SCS is an ordinal scale where the subject responds to the question, "On a 0 to 10 scale, if 0 represents the most uncomfortable socket fit you can imagine, and 10 represents the most comfortable socket fit, how would you score the comfort of the socket of your artificial limb at the moment?"
Time Frame: 7 weeks
Population: Cross-sectional analysis was conducted with the 19 participants who completed the 7-week data collection visit for this outcome measure for each socket.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- NU-FlexSIV Socket: Participants wore the NU-FlexSIV Socket for 7 weeks
- Ischial Containment Socket: Participants wore the Ischial Containment Socket for 7 weeks
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
score on a scale | 8.5 (1.1) | 6.8 (1.8)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p < 0.001, t-test, 2 sided — alpha = 0.05; paired t-test; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.8 to 2.3], Standard Deviation 1.5

2. Secondary Outcome: Walking Speed Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: Walking speed was assessed after each socket was worn for 7 weeks. Participants walked along a 12 meter, level walkway at their normal self-selected speed. Marker based motion capture was used to assess walking speed (m/s).
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- NU-FlexSIV Socket: Participant wore the NU-FlexSIV Socket for 7 weeks.
- Ischial Containment Socket: Participant wore the Ischial Containment Socket for 7 weeks.
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
m/s | 1.14 (0.20) | 1.13 (0.17)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.664, t-test, 2 sided — p-value was adjusted using a Bonferonni correction with alpha set at 0.017; paired t-test; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.04], Standard Deviation 0.1

3. Secondary Outcome: Step Length Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: Step length was assessed after each socket was worn for 7 weeks. Participants walked along a 12 meter, level walkway at their normal self-selected speed. Marker based motion capture was used to assess step length (cm).
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
cm | 70.26 (10.20) | 68.56 (9.63)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.026, t-test, 2 sided — p-value was adjusted using a Bonferonni correction with alpha set at 0.017; paired t-test; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-3.17 to -0.23], Standard Deviation 3.05

4. Secondary Outcome: Hip Extension Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: Hip extension was assessed after each socket was worn for 7 weeks. Participants walked along a 12 meter, level walkway at their normal self-selected speed. Marker based motion capture was used to assess hip extension (degrees).
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
degrees | -3.30 (8.65) | -3.10 (8.67)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.847, t-test, 2 sided — p-value was adjusted using a Bonferonni correction with alpha set at 0.025; paired t-test; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-2 to 2.42], Standard Deviation 4.58

5. Secondary Outcome: Hip Range of Motion Between the IC Socket and NU-FlexSIV Socket 7 Weeks.
Description: Hip range of motion was assessed after each socket was worn for 7 weeks. Participants walked along a 12 meter, level walkway at their normal self-selected speed. Marker based motion capture was used to assess hip range of motion (degrees).
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
degrees | 44.34 (4.90) | 43.30 (5.22)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p < 0.017, t-test, 2 sided — p-value was adjusted using a Bonferonni correction with alpha set at 0.017; paired t-test; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-2.42 to 0.34], Standard Deviation 2.87

6. Secondary Outcome: Trunk Motion Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: Trunk motion was assessed after each socket was worn for 7 weeks. Participants walked along a 12 meter, level walkway at their normal self-selected speed. Marker based motion capture was used to assess trunk motion (degrees).
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
degrees | 3.61 (3.23) | 3.73 (3.70)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Other; p = 0.7, t-test, 2 sided — p-value was adjusted using a Bonferonni correction with alpha set at 0.025; paired t-test; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.53 to 0.77], Standard Deviation 4.58

7. Secondary Outcome: Orthotics and Prosthetics Users' Survey (OPUS) Lower-Extremity Functional Status Measure Between the IC Socket and NU-FlexSIV Socket at 7 Weeks
Description: Lower-Extremity Functional Status was assessed after each socket was worn for 7 weeks. The OPUS Lower-Extremity Functional Status measure is a self-report instrument that assesses functional status in persons who use orthoses and prostheses. It is comprised of 20 items rated on a 5-point rating scale. Responses to items are summed to produce a total score for the measure (0 to 80) with higher scores representing better functional status.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
score on a scale | 58.3 (10.4) | 55.5 (13.9)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.20, t-test, 2 sided — alpha = 0.05; paired t-test; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-1.6 to 7.0], Standard Deviation 8.9

8. Secondary Outcome: Orthotics andProsthetics Users' Survey (OPUS) Health Related Quality of Life Index Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: Health Related Quality of life was assessed after each socket was worn for 7 weeks. The OPUS Health Related Quality of Life measure is self-report instrument comprised of 23 items that are evaluated with a 5-point rating scale. Responses to items are summed to produce a total score for the index (0 to 92) with higher scores representing better quality of life.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
score on a scale | 69.1 (17.1) | 70.2 (16.3)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.62, t-test, 2 sided — alpha = 0.05; paired t-test; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-6.0 to 3.7], Standard Deviation 10

9. Secondary Outcome: Orthotics and Prosthetics Users' Survey (OPUS) Satisfaction With Device Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: Satisfaction with Device was assessed after each socket was worn for 7 weeks. The OPUS Satisfaction with Device measure is a set of 11 items rated on a 5-point rating scale. Responses to items are summed to produce a total score. 9 items were used in this study for a possible score of 9 to 45 with higher scores representing better satisfaction.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
score on a scale | 35.1 (6.5) | 32.5 (7.3)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.07, t-test, 2 sided — alpha = 0.05; paired t-test; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-0.2 to 5.3], Standard Deviation 5.7

10. Secondary Outcome: 5-Times Rapid Sit-to-Stand Test (RSTS) Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: The 5-Times Rapid-Sit-to-Stand Test was assessed after each socket was worn for 7 weeks. Participants were asked to rise from a chair of standard height five times as fast as possible with their arms folded across their chests. Performance was timed.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 17 | 17
seconds | 12.7 (4.5) | 14.8 (8.8)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.18, t-test, 2 sided — alpha = 0.05; paired t-test; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-5.4 to 1.1], Standard Deviation 6.3

11. Secondary Outcome: Four-Square-Step Test (FSST) Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: The Four-Square-Step Test was assessed after each socket was worn for 7 weeks. Four sticks were placed flat on the floor in a cross that denoted a square. Participants were asked to complete a stepping sequence as fast as possible. Performance was timed.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- IC Socket: Participants wore the Ischial Containment Socket for 7 weeks.
Arm/Group | NU-FlexSIV Socket | IC Socket
Number analyzed (Participants) | 19 | 19
seconds | 9.7 (2.0) | 9.5 (2.1)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs IC Socket; Test type: Superiority; p = 0.47, t-test, 2 sided — alpha = 0.05; paired t-test; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.9], Standard Deviation 1.3

12. Secondary Outcome: T-Test of Agility (T-Test) Between the IC Socket and NU-FlexSIV Socket at 7 Weeks.
Description: The T-Test was assessed after each socket was worn for 7 weeks. Four markers were set out so a "T" could be traced among them. The subject was asked to move as fast as possible between the markers, moving forwards, sideways and backwards. Performance was timed and reported in seconds.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: seconds
Arm/Group | NU-FlexSIV Socket | Ischial Containment Socket
Number analyzed (Participants) | 19 | 19
seconds | 41.8 (13.3) | 41.4 (12.4)
Statistical Analysis 1: Comparison: NU-FlexSIV Socket vs Ischial Containment Socket; Test type: Superiority; p = 0.68, t-test, 2 sided — alpha = 0.05; paired t-test; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.4 to 2.0], Standard Deviation 3.5

ADVERSE EVENTS:
Time Frame: 7 weeks for each intervention.
Arm/Group | Ischial Containment Socket | NU-FlexSIV Socket
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 14/25 | 18/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ischial Containment Socket (N=25) | NU-FlexSIV Socket (N=25)
residual limb skin issue (Injury, poisoning and procedural complications) | 7 (7) | 9 (9) — residual limb itching, skin reaction, blister or sore
fall during testing (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
low back pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
prosthetic foot came loose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
residual limb volume changes (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
muscle soreness or cramping (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
socket caused pain/discomfort (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02678247/Prot_SAP_000.pdf